CLINICAL TRIAL: NCT03323554
Title: Prospective Interventional Safety and Efficacy Study of USTRAP™ in Male Urinary Incontinence. an Open, Randomised, Multicentre Study Versus Artificial Sphincter.
Brief Title: Safety and Efficacy Study of USTRAP™ in Male Urinary Incontinence
Acronym: PROSPECT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Quanta Medical (Industry)
Collaborators: Cousin Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2782
Record Dates: First submitted 2017-10-24; First posted 2017-10-27 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-07

CONDITIONS: Urinary Incontinence
Keywords: radical prostatectomy , Device,
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Intervention Model Description: a prospective, randomised, multicentre, comparative, open label, non-inferiority study in parallel groups of patients presenting stress urinary incontinence following prostate ablation for cancer.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ustrap® (Experimental): Ustrap is a new adjustable-pressure 4-arm device
  Interventions: Device: Ustrap®
- AMS 800® (Active Comparator): Artificial sphincter currently considered the gold standard device in this field
  Interventions: Device: AMS 800®

INTERVENTIONS:
Device: Ustrap® — Patients will receive Ustrap® under general or loco-regional anaesthesia, by perineal approach.
  Arms: Ustrap®
Device: AMS 800® — Patients will receive AMS 800® under general or loco-regional anaesthesia. Small openings are made near the scrotum and below the abdomen to insert an inflatable cuff, a pump and a small balloon (pressure regulating balloon).
  Arms: AMS 800®

SUMMARY:
Few surgical methods to treat male stress urinary incontinence have been assessed in comparative, randomised interventional studies.

Ustrap is a new adjustable-pressure 4-arm device. The artificial sphincter is currently considered the gold standard device in this field.

The aim of this randomised prospective international study is to assess the efficacy and safety of the Ustrap® device comparatively with an artificial sphincter (AMS800) in the treatment of stress urinary incontinence following prostate removal in cancer patients.

ELIGIBILITY:
Inclusion Criteria:

Disease-related criteria:

* persistent urinary incontinence >= 12 months following radical prostatectomy for prostate adenocarcinoma
* presenting an indication for surgical insertion of a medical device
* 24h PAD test > 100 g per day
* controlled prostate adenocarcinoma, with PSA ≤ 1 ng/ml

Population-related criteria:

* male subjects aged 18 years and over
* having provided free, informed written consent to take part in the study
* patients independent and able to use the collar without difficulty and able to manage an artificial sphincter
* Patient able to understand and sign the consent form and to complete questionnaires
* Patient without mental impairment
* Patients belonging to or covered by Social Security.

Exclusion Criteria:

Disease-related criteria:

* Documented neurological bladder or history of neurological disease liable to interfere with urinary symptoms.
* Presence of urethral anastomotic stenosis preventing passage of the fiberscope at the initial endoscopy
* Severe symptomatic hyperactive or hypoactive bladder not controlled by drug therapy
* Severe constitutional haemorrhagic disease or haemophilia
* Patients presenting urinary infection not controlled
* Patients presenting severe renal failure and obstructive pathologies of the upper urinary tract with severe renal failure.
* Patients presenting deep immune deficiency
* Patient presenting recto-urethral fistula
* Patient with tumor of bladder
* Patient having bladder stones with failure of bladder stone treatment

Criteria related to incontinence treatment:

* Allergy to any of the components of the medical devices
* History of surgery to insert a medical device for treatment of incontinence (e.g. artificial sphincter, suburethral strap, continence balloons, etc.)
* History of periurethral injection of filling agents
* Inability to use either of the study devices
* Drug treatment: duloxetine or any treatment likely to modify continence results
* Not receiving and not likely to receive radiotherapy at any time throughout the 12-month follow-up period Population-related criteria
* Foreseeable unavailability during the study . Patient deprived of liberty by administrative or judicial decision or under legal guardianship
* Participation in another clinical trial in the 3 months preceding the initial visit

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
comparison of succes rate | 12 months
  Succes being defined as the absence of use of protective pads, or in the case of use of safety protection comprising a test PAD over 24h, wet weight indicating collection of ≤ 10 g liquid, and the absence of corrective surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Charles Nicolle, Rouen, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Herschorn S, Bruschini H, Comiter C, Grise P, Hanus T, Kirschner-Hermanns R, Abrams P; Committee of the International Consultation on Incontinence. Surgical treatment of stress incontinence in men. Neurourol Urodyn. 2010;29(1):179-90. doi: 10.1002/nau.20844. PMID 20025026
- See also: Related Info — http://uroweb.org/guideline/urinary-incontinence
- See also: Related Info — https://doi.org/10.1016/S1569-9056(16)60199-9